CLINICAL TRIAL: NCT06762899
Title: Effect of Chronic Mechanical Neck Pain on Isokinetic Characteristics of Rotator Cuff Muscles in Adults
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Adel Mohamed Hegazy, demonstrator, Cairo University
Other Study IDs: P.T.REC/012/005142
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Chronic Mechanical Neck Pain
Keywords: Isokinetic; Mechanical neck pain; Neuromuscular; Rotator cuff; Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- chronic mechanical neck pain group: chronic mechanical neck pain was assessed by visual analogue scale to determine pain intensity and neck disability index to determine level of disability caused by neck pain isokinetic characteristics of rotator cuff muscles were assessed by biodex isokinetic dynamometer

SUMMARY:
Statement of the problem:Would chronic mechanical neck pain affect isokinetic characteristics of Rotator Cuff muscles in adults? it was assumed that There would be no significant effect of chronic mechanical neck pain on isokinetic characteristics of Rotator Cuff muscles in adults.

DETAILED DESCRIPTION:
Sixty-six participants of both sexes between (18 and 29 years old) were enrolled in this study. Thirty-three participants with Chronic Mechanical Neck Pain(CMNP) , thirty-three participants without CMNP. They were recruited from out-patient clinics of faculty of physical therapy, Cairo University.

instrumentation :neck pain intensity was determined by visual analogue scale , neck pain intensity was determined by neck disability index , isokinetic characteristics of rotator cuff muscles was determined by biodex isokinetic dynamometer .

ELIGIBILITY:
Inclusion Criteria:

Subjects were included according to the following criteria:

* Thirty-three participants with Chronic Mechanical Neck Pain(CMNP) and Thirty-three healthy participants would be assigned into two groups; healthy control group (A) and CMNP group (B).
* Right and left- handed subjects.
* Both sexes between 18-29 years old
* (0-4 mm) no pain, (5-44 mm) mild pain, (45-74 mm) moderate pain, (75-100 mm) severe neck pain on visual analogue scale .
* Chronic neck pain > 12 weeks .
* They did not take any painkillers for the last 48 hours before assessment.

Exclusion criteria:

Subjects were excluded if they have any of the following:

* Shoulder-related pain.
* The existence of any anomalies in the neck and shoulder areas.
* A history of trauma or severe illnesses such as diabetes, cancer, fibromyalgia, or any kind of tumor.
* Disc herniation; history of identifiable structural injury.
* Past incidents of whiplash injury.
* Prior surgery; fractures.
* Pregnancy.
* Any prior rehabilitative therapy received during the last three months.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sixty-six participants of both sexes between (18 and 29 years old) were enrolled in this study.Thirty-three participants with CMNP, thirty-three participants without CMNP.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
isokinetic characteristics of rotator cuff muscles were assessed by biodex isokinetic dynamometer | baseline only

CONTACTS AND LOCATIONS:
Overall Officials: sohair shehata rezk allah, professor, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of Physical Therapy ,Cairo University, Cairo
  - Out Patient Clinic of Faculty of Physical Therapy , Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided